CLINICAL TRIAL: NCT00621270
Title: A 6-Week Randomised Double-Blind, Placebo-Controlled Study of BCI-540 80 mg q.d. and 80 mg t.i.d. in the Treatment of Adults With Major Depressive Disorder and Concomitant Anxiety
Brief Title: Safety and Effectiveness Study of BCI-540 Versus Placebo in the Treatment of Major Depressive Disorder With Concomitant Anxiety
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BrainCells Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BCI-540-CL-001
Record Dates: First submitted 2008-02-11; First posted 2008-02-22 (Estimated); Last update posted 2011-10-24 (Estimated); Status verified 2011-10

CONDITIONS: Major Depressive Disorder; Anxiety
Keywords: Major Depression Neurogenesis; Major Depressive Disorder with Concomitant Anxiety
MeSH Terms: conditions — Depressive Disorder, Major; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): BCI-540 80 mg once a day (q.d.)
  Interventions: Drug: BCI-540
- 2 (Experimental): BCI-540 80 mg three times a day (t.i.d.)
  Interventions: Drug: BCI-540
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: BCI-540

INTERVENTIONS:
Drug: BCI-540 — BCI-540 80 mg once (q.d.) or three times (t.i.d.) a day versus placebo

SUMMARY:
The purpose of this study is to determine whether BCI-540 80 mg given once daily (q.d.) or three times daily (t.i.d.) is effective in the treatment of major depression with concomitant anxiety.

DETAILED DESCRIPTION:
BCI-540 has been shown to be neurogenic in the Sponsor's in vitro neural stem cell analyses and in vivo animal models of depression and anxiety. These observations and the recent findings linking hippocampal function and neurogenesis to mood disorders support the evaluation of the efficacy, safety, and tolerability of BCI-540 in patients with major depressive disorder with concomitant anxiety.

ELIGIBILITY:
Inclusion Criteria:

* The patient meets the DSM IV-TR criteria for Major Depressive Disorder (MDD) as determined by the Mini-International Neuropsychiatric Interview (MINI) and psychiatric evaluation.
* The patient has a score of 20 or more on the HAM D17 scale, a score of 30 or more on the IDS-C30 and a score of 15 or more on the HAM-A scale at the Screening and Baseline visits.
* The patient has a score of at least 2 on items 1 and 2 of the HAM-A scale at the Screening and Baseline visits.
* The patient has a Clinical Global Impression of Severity (CGI S) rating of 4 or higher at the Screening and Baseline visits.
* The patient has recurrent MDD.
* The patient did not respond to at least one but no more than five adequate antidepressant trials during the current MDD episode.
* The patient is living with another adult or has daily contact with an adult and contact information for the patient and this adult is available to the investigator.
* Female patients of childbearing potential must be using a reliable, medically acceptable form of contraception for at least 30 days prior to the screening visit and must agree to continue such use throughout the duration of the study and for 30 days after the final dose of study drug.

Exclusion Criteria:

* The patient has a decrease of 20% or more in HAM D17 total score or HAM-A total score from the screening visit to the Baseline visit.
* The patient represents significant risk of suicide in the opinion of the investigator at the screening or Baseline visit.
* The patient has any other psychiatric Axis-I disorder (except GAD) as a principal diagnosis within 6 months of Screening.
* The patient has a history of obsessive compulsive disorder, psychotic disorder, bipolar disorder, mental retardation.
* The patient has a history of alcohol or substance (excluding nicotine or caffeine) abuse within 3 months of the screening visit, alcohol or substance dependence within 6 months of Screening.
* The patient shows current evidence of substance abuse confirmed by results of a urine drug screen.
* The patient has used an antidepressant medication (SSRI/SNRI or any other antidepressant medication, including MAOIs), within 1 week of Baseline(fluoxetine within 5 weeks).
* The patient has a history of low RBC count, low hemoglobin, low WBC count, low platelets, or low reticulocyte counts of any aetiology other than that known to be related to blood loss, iron deficiency, or pregnancy.
* The patient shows current evidence of macrocytosis, low RBC count, low haemoglobin, low WBC count, or low platelet count of any aetiology.
* The patient will use drugs during the study (including follow-up) that are known to be related to agranulocytosis and/or aplastic anaemia.
* The patient will receive interpersonal therapy and/or short-term (brief) dynamic therapy during the study.
* The patient received ECT within 3 months of Screening.
* The patient received depot antipsychotic therapy at any time.
* The patient has used any antipsychotic or anxiolytic medications within 1 week of Screening.
* The patient has used any drugs with known psychotropic properties or any non-psychotropic drugs with potential CNS effects within one week or 5-half lives (whichever is longer) of Screening.
* The patient has a clinically significant cardiovascular, endocrine, hepatic, renal, pulmonary, gastrointestinal, neurological, malignancy, metabolic, psychiatric or other condition that might be detrimental to the patient if he or she participates in the study.
* The patient has a known hypersensitivity to any cholinesterase inhibitors or cholinergic agonist drugs.
* The patient is a pregnant or lactating woman.
* The patient has a history of seizures.
* The patient has clinically significant abnormalities on screening physical examination, ECG, serum chemistry, urinalysis tests, including thyroid stimulating hormone levels, as judged by the investigator.
* The patient has a known positivity for human immunodeficiency virus, hepatitis B surface-antigen, or hepatitis C virus antibody.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 115 (Actual)
Dates: Start 2008-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Co-primary outcome measures will be the change from Baseline to Week 6 on the total score of the Inventory of Depressive Symptomatology-Clinician Version (IDS-C30) and the Hamilton Rating Scale for Anxiety (HAM-A). | Week 6

SECONDARY OUTCOMES:
The safety, tolerability and side effect profile of BCI-540 will also be measured by adverse events, clinical laboratory values, electrocardiograms, vital signs, and the Physician Withdrawal Checklist (PWC). | Weeks 2, 4, 6, 7 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Allan H. Young, MB ChB, MPhil, PhD, FRCPsych, Study Chair — Institute of Mental Health, Dept. of Psychiatry, University of British Columbia
Locations (16):
- Canada (16):
  - Grey Nuns Hospital, Clinical Research, Edmonton, Alberta
  - Okanagan Clinical Trials, Kelowna, British Columbia
  - Dr. Alexander McIntyre, Inc, Penticton, British Columbia
  - University of British Columbia Mood Disorders Centre, Vancouver, British Columbia
  - Dr. D. McIntosh & Dr. K. Kjernisted Clinical Research Inc., Vancouver, British Columbia
  - Eden Mental Health Centre, Winkler, Manitoba
  - Sanjay Siddhartha, MD, Miramichi, New Brunswick
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Autar K. Munshi, MD, Sydney, Nova Scotia
  - Robert Fairbairn, MD, Chatham, Ontario
  - Providence Care Mental Health Services, Kingston, Ontario
  - Robert G. Luton, MD, London, Ontario
  - Anxiety and Mood Disorder Center, Mississauga, Ontario
  - Ottawa Psychopharmacology Clinic, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network, Dept. of Psychiatry, Toronto, Ontario